CLINICAL TRIAL: NCT03156023
Title: A Randomized, Double Blind Placebo Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Subcutaneous Doses of AMG 570 in Subjects With Rheumatoid Arthritis
Brief Title: Multiple Ascending Doses of Rozibafusp Alfa (AMG 570) in Adults With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150196; 2017-000337-31 (EudraCT Number)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — rozibafusp alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rozibafusp Alfa (Experimental): Participants will receive rozibafusp alfa administered subcutaneously once every 2 weeks for up to 10 weeks (6 doses). Rozibafusp alfa doses will range from 70 to 420 mg.
  Escalation to a higher dose cohort will be contingent on a review indicating that the previous dose regimen has been found to demonstrate an acceptable safety and tolerability profile at a dose level review meeting (DLRM).
  Interventions: Drug: Rozibafusp Alfa
- Placebo (Placebo Comparator): Participants will receive matching placebo to rozibafusp alfa administered subcutaneously once every 2 weeks for up to 10 weeks (6 doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rozibafusp Alfa — Administered by subcutaneous injection once every 2 weeks.
  Other Names: AMG 570
  Arms: Rozibafusp Alfa
Drug: Placebo — Administered by subcutaneous injection once every 2 weeks.
  Arms: Placebo

SUMMARY:
A study to evaluate safety and tolerability and characterize the pharmacokinetic (PK) profile of rozibafusp alfa following multiple dose administration in adults with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 18-35 kg/m^2
* Diagnosed with RA (disease duration of at least 6 months)
* Stable dose of methotrexate (5-25 mg weekly for ≥ 4 weeks)
* Immunizations up to date
* Willing to use highly effective contraception during treatment and through end-of-study

Exclusion Criteria:

* Uncontrolled, clinically significant systemic disease other than RA (i.e., diabetes mellitus, liver disease, asthma, cardiovascular disease, hypertension)
* Malignancy within 5 years
* Presence of serious infection, recurrent/chronic infections
* Class IV RA according to American College of Rheumatology/ (ACR) revised response criteria
* Diagnosed with Felty's syndrome
* Known or suspected sensitivity to mammalian cell-derived products
* History of alcohol and/or substance abuse within the last 12 months
* Receipt of rituximab at any time in the past
* Evidence of renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (3):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
- Charite Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Abuqayyas L, Chen PW, Dos Santos MT, Parnes JR, Doshi S, Dutta S, Houk BE. Pharmacokinetics and Pharmacokinetic/Pharmacodynamic Properties of Rozibafusp Alfa, a Bispecific Inhibitor of BAFF and ICOSL: Analyses of Phase I Clinical Trials. Clin Pharmacol Ther. 2023 Aug;114(2):371-380. doi: 10.1002/cpt.2929. Epub 2023 May 24. PMID 37150935
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 centers in the United States and Germany. Participants with rheumatoid arthritis were enrolled from 14 August 2017 to 20 February 2019.
Pre-assignment Details: The study consisted of 4 multiple ascending dose cohorts. Within each cohort participants were randomized in a 3:1 ratio to receive rozibafusp alfa or placebo. Escalation to a higher dose cohort was contingent on a review to confirm that the previous dose regimen(s) demonstrated an acceptable safety and tolerability profile.
Groups:
- Placebo: Participants received placebo administered by subcutaneous injection once every 2 weeks for 10 weeks (6 doses).
- Rozibafusp Alfa 70 mg: Participants received 70 mg rozibafusp alfa administered by subcutaneous injection once every 2 weeks for 10 weeks (6 doses).
- Rozibafusp Alfa 140 mg: Participants received 140 mg rozibafusp alfa administered by subcutaneous injection once every 2 weeks for 10 weeks (6 doses).
- Rozibafusp Alfa 210 mg: Participants received 210 mg rozibafusp alfa administered by subcutaneous injection once every 2 weeks for 10 weeks (6 doses).
- Rozibafusp Alfa 420 mg: Participants received 420 mg rozibafusp alfa administered by subcutaneous injection once every 2 weeks for 10 weeks (6 doses).
Period: Overall Study
Arm/Group | Placebo | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Started | 8 | 7 | 6 | 6 | 7
Completed | 7 | 7 | 4 | 5 | 5
Not Completed | 1 | 0 | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of rozibafusp alfa or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg | Total
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 7 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (8.6) | 60.4 (11.9) | 61.0 (11.2) | 60.7 (9.6) | 58.7 (4.9) | 60.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 4 | 6 | 5 | 28
  Male | 2 | 0 | 2 | 0 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 7 | 6 | 5 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2
  White | 7 | 7 | 5 | 6 | 7 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial subject, including worsening of a pre-existing medical condition and clinically significant changes in laboratory test results and physical exam findings. The event does not necessarily have a causal relationship with study treatment.
  AEs were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4, where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe or medically significant, Grade 4 = Life-threatening, and Grade 5 = Death.
  A serious adverse event is defined as an AE that met at least 1 of the following serious criteria:
  * fatal;
  * life threatening;
  * required in patient hospitalization or prolongation of existing hospitalization;
  * resulted in persistent or significant disability/incapacity;
  * congenital anomaly/birth defect;
  * other medically important serious event. The investigator assessed whether each AE was related to study drug.
Time Frame: From first dose of study drug to 24 weeks after last dose (up to 34 weeks).
Population: All randomized participants who received at least 1 dose of rozibafusp alfa or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 8 | 7 | 6 | 6 | 7
Participants
  Any treatment-emergent adverse event (TEAE) | 7 | 6 | 6 | 6 | 7
  TEAE Grade ≥ 2 | 4 | 5 | 3 | 4 | 6
  TEAE Grade ≥ 3 | 0 | 1 | 1 | 0 | 0
  TEAE Grade ≥ 4 | 0 | 0 | 0 | 0 | 0
  Serious adverse events | 0 | 1 | 1 | 0 | 0
  TEAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0
  Severe adverse events | 0 | 1 | 1 | 0 | 0
  Life-threatening adverse events | 0 | 0 | 0 | 0 | 0
  Fatal adverse events | 0.0 | 0 | 0 | 0 | 0
  Treatment-related TEAE (TRAE) | 2 | 0 | 1 | 1 | 4
  TRAE Grade ≥ 2 | 2 | 0 | 0 | 1 | 2
  TRAE Grade ≥ 3 | 0 | 0 | 0 | 0 | 0
  TRAE Grade ≥ 4 | 0 | 0 | 0 | 0 | 0
  Treatment-related serious adverse events | 0 | 0 | 0 | 0 | 0
  TRAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0
  Severe TRAE | 0 | 0 | 0 | 0 | 0
  Life-threatening TRAE | 0 | 0 | 0 | 0 | 0
  Fatal TRAE | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Rozibafusp Alfa
Time Frame: Day 1 predose and 6, 12, 24, 48, 72, 144, 168, and 336 hours post-dose. Week 10 predose and 6, 12, 24, 48, 72, 144, 168, and 336 hours and at 3, 4, 5, 6, 8, 10, and 12 weeks post-dose.
Population: The pharmacokinetic (PK) parameter analysis set includes all randomized participants who received rozibafusp alfa and for whom PK parameters were adequately estimated.
Measure: Median (Full Range); unit: days
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 7 | 6 | 6 | 7
days
  Day 1 | 3.0 [3.0 to 7.0] | 3.0 [2.0 to 6.0] | 4.5 [3.0 to 7.0] | 6.0 [3.0 to 6.1]
  Week 10: number analyzed (Participants) | 7 | 4 | 6 | 6
  Week 10 | 3.0 [3.0 to 7.0] | 5.0 [2.0 to 7.0] | 2.5 [2.0 to 3.0] | 2.5 [0.98 to 8.1]

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Rozibafusp Alfa
Time Frame: as for outcome 2
Population: PK parameter analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 7 | 6 | 6 | 7
μg/mL
  Day 1 | 2.56 (1.51) | 8.34 (4.09) | 13.7 (7.22) | 24.1 (11.1)
  Week 10: number analyzed (Participants) | 7 | 4 | 6 | 6
  Week 10 | 6.85 (4.59) | 22.7 (12.6) | 44.1 (13.4) | 67.9 (18.7)

4. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 14 Days Postdose (AUC0-tau) for Rozibafusp Alfa
Time Frame: Day 1 predose and 6, 12, 24, 48, 72, 144, 168, and 336 hours post-dose. Week 10 predose and 6, 12, 24, 48, 72, 144, 168, and 336 hours post-dose.
Population: PK parameter analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 7 | 6 | 6 | 5
day*μg/mL
  Day 1: number analyzed (Participants) | 7 | 6 | 5 | 5
  Day 1 | 22.6 (14.7) | 86.2 (47.1) | 143 (85.3) | 265 (162)
  Week 10: number analyzed (Participants) | 7 | 4 | 6 | 5
  Week 10 | 57.1 (33.6) | 284 (170) | 510 (151) | 864 (206)

5. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) for Rozibafusp Alfa
Time Frame: Week 10 predose and 6, 12, 24, 48, 72, 144, 168, and 336 hours and at 3, 4, 5, 6, 8, 10, and 12 weeks post-dose.
Population: PK parameter analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 6 | 4 | 6 | 5
day*μg/mL | 107 (82.4) | 651 (483) | 1110 (447) | 2160 (606)

6. Secondary Outcome: Terminal Half-life of Rozibafusp Alfa
Time Frame: Week 10 predose and 6, 12, 24, 48, 72, 144, 168, and 336 hours and at 3, 4, 5, 6, 8, 10, and 12 weeks post-dose.
Population: PK parameter analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 6 | 4 | 6 | 5
days | 4.62 (1.05) | 5.62 (1.14) | 6.68 (3.48) | 9.50 (3.44)

7. Secondary Outcome: Accumulation Ratio of AUCtau
Description: Accumulation ratio is the ratio of AUCtau after the last dosing interval (week 10) divided by AUCtau after the first dosing interval (day 1).
Time Frame: as for outcome 4
Population: PK parameter analysis set with available AUCtau data at day 1 and week 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 7 | 4 | 5 | 4
ratio | 2.94 (1.75) | 3.55 (1.20) | 4.41 (2.28) | 4.27 (3.24)

8. Secondary Outcome: Accumulation Ratio of Cmax
Description: Accumulation ratio is the ratio of Cmax after the last dosing interval (week 10) divided by Cmax after the first dosing interval (day 1).
Time Frame: as for outcome 4
Population: PK parameter analysis set with available Cmax data at day 1 and week 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
Number analyzed (Participants) | 7 | 4 | 6 | 6
ratio | 3.08 (1.96) | 3.00 (1.05) | 4.06 (2.12) | 3.71 (2.38)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 24 weeks after last dose (up to 34 weeks).
Arm/Group | Placebo | Rozibafusp Alfa 70 mg | Rozibafusp Alfa 140 mg | Rozibafusp Alfa 210 mg | Rozibafusp Alfa 420 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/7 | 1/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 7/8 | 6/7 | 6/6 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Rozibafusp Alfa 70 mg (N=7) | Rozibafusp Alfa 140 mg (N=6) | Rozibafusp Alfa 210 mg (N=6) | Rozibafusp Alfa 420 mg (N=7)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Rozibafusp Alfa 70 mg (N=7) | Rozibafusp Alfa 140 mg (N=6) | Rozibafusp Alfa 210 mg (N=6) | Rozibafusp Alfa 420 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 2 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Mycoplasma infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 2
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT03156023/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03156023/SAP_001.pdf